CLINICAL TRIAL: NCT04639804
Title: An Open-label, Randomized, Crossover Study to Evaluate the Pharmacokinetic Interaction Between Tegoprazan and Non-steroidal Anti-inflammatory Drugs (NSAIDs) After Multiple Oral Dosing in Healthy Male Volunteers
Brief Title: Pharmacokinetic Interaction Between Tegoprazan and NSAIDs After Multiple Oral Dosing in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IN_APA_117
Record Dates: First submitted 2020-11-16; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: drug-drug interaction; pharmacokinetic
MeSH Terms: interventions — tegoprazan; Naproxen; aceclofenac; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tegoprazan 50 mg (Active Comparator): Multiple doses of tegoprazan alone once daily (QD) for 7 days
  Interventions: Drug: Tegoprazan
- NSAIDs (Active Comparator): Multiple doses of NSAIDs alone twice daily (BID) for 7 days
  Interventions: Drug: Naproxen; Drug: Aceclofenac; Drug: Celecoxib
- Tegoprazan 50 mg + NSAIDs (Active Comparator): Multiple doses of tegoprazan QD in combination with NSAIDs BID for 7 days
  Interventions: Drug: Tegoprazan; Drug: Naproxen; Drug: Aceclofenac; Drug: Celecoxib

INTERVENTIONS:
Drug: Tegoprazan — Tegoprazan 50 mg tablet
  Other Names: K-CAB
  Arms: Tegoprazan 50 mg; Tegoprazan 50 mg + NSAIDs
Drug: Naproxen — Naproxen 500 mg tablet
  Other Names: Naxen-F
  Arms: NSAIDs; Tegoprazan 50 mg + NSAIDs
Drug: Aceclofenac — Aceclofenac 100 mg tablet
  Other Names: Airtal
  Arms: NSAIDs; Tegoprazan 50 mg + NSAIDs
Drug: Celecoxib — Celecoxib 200 mg capsule
  Other Names: Celebrex 200 mg
  Arms: NSAIDs; Tegoprazan 50 mg + NSAIDs

SUMMARY:
This study aims to evaluate the pharmacokinetic (PK) interaction between tegoprazan and non-steroidal anti-inflammatory drugs (NSAIDs) after given each alone and in their combination in healthy male adults.

DETAILED DESCRIPTION:
A randomized, open-label, multiple-dose, 6-sequence-arm, 3-period cross-over study

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged ≥ 19 and < 55 year-old at screening
* Body mass index (BMI) ≥ 19.0 kg/m2 and < 27.0 kg/m2 with a body weight ≥ 55 kg at screening.

Exclusion Criteria:

* History or evidence of clinically significant disease
* History of GI disease or surgery that may affect the absorption of a drug
* Laboratory test result which falls into the following values( ALT or AST > 2 × upper limit of normal (ULN))
* History of regular alcohol consumption exceeding 210 g/week within 6 months
* Daily use of ≥ 20 cigarettes within 6 months
* Has taken any investigational agent within 6 months prior to the first dose of IMP
* Subjects who are considered ineligible to participate in this study at the discretion of the investigator.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2020-07-26 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
AUCτ of tegoprazan and NSAIDs | pre-dose (0 hour) on Day1, Day5, Day6 and pre-dose up to 24 hours post-dose on Day7
  Area under the plasma concentration-time curve during a steady-state dosing interval (τ) of tegoprazan and NSAIDs
Css,max of tegoprazan and NSAIDs | pre-dose (0 hour) on Day1, Day5, Day6 and pre-dose up to 24 hours post-dose on Day7
  Maximum Plasma Concentration at Steady State of tegoprazan and NSAIDs

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, MD, PhD, Principal Investigator — Chonbuk university hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

REFERENCES:
- [Derived] Moon SJ, Shin N, Kang M, Kim B, Kim MG. Pharmacokinetic Interactions Between Tegoprazan and Naproxen, Aceclofenac, and Celecoxib in Healthy Korean Male Subjects. Clin Ther. 2022 Jul;44(7):930-944.e1. doi: 10.1016/j.clinthera.2022.06.002. Epub 2022 Jul 1. PMID 35787943